CLINICAL TRIAL: NCT06852963
Title: A Repeat-Dose, Open-Label, Two Arm Safety and Efficacy Study of Two Doses of VP-001 (30 μg and 75 μg) Administered Intravitreally in Participants With Confirmed PRPF31 Mutation-Associated Retinal Dystrophy, Including Participants Previously Treated With VP001 in the PLATYPUS Study (Protocol # VP001-101) or WALLABY Study (Protocol # VP001-102) for a Minimum of 8 Weeks
Brief Title: A Repeat-Dose, Open-Label, Two Arm Safety and Efficacy Study of Two Doses of VP-001 Administered Intravitreally in Participants With Confirmed PRPF31 Mutation-Associated Retinal Dystrophy, Including Participants Previously Treated With VP001
Acronym: DINGO
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PYC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VP001-CL103
Record Dates: First submitted 2025-02-20; First posted 2025-02-28 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-03

CONDITIONS: Retinitis Pigmentosa 11; Retinal Degeneration; Retinal Disease; Eye Diseases Hereditary; Retinal Dystrophies
Keywords: VP-001-CL103
MeSH Terms: conditions — Retinitis Pigmentosa 11; Retinal Degeneration; Retinal Diseases; Eye Diseases, Hereditary; Retinal Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: 30ug VP-001 every 8 weeks (Experimental)
  Interventions: Drug: VP-001
- Cohort 2: 75ug of VP-001 every 12 weeks (Experimental)
  Interventions: Drug: VP-001

INTERVENTIONS:
Drug: VP-001 — VP-001 is an oligonucleotide-peptide conjugate administered intravitreally.

SUMMARY:
This is a Phase 1/2 repeat-dose, open-label, two-arm, parallel group safety and efficacy study of two doses of VP-001 (30 μg and 75 μg) in participants with confirmed PRPF31 mutation-associated retinal dystrophy, including participants previously treated with VP001 in the PLATYPUS Study or WALLABY Study for a minimum of 8 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female sex; ≥18 years of age at Day 1/Baseline (Visit 2)
* May have been previously enrolled in PLATYPUS Part B (Protocol #VP001-CL101) or WALLABY (Protocol #VP001-CL102) study. At Screening Visit in this study, participants must have completed at least 8 weeks after last study agent administration in PLATYPUS Part B (Protocol #VP001-CL101) or WALLABY (Protocol # VP001-CL102) study
* Have a confirmed clinical diagnosis of Retinitis Pigmentosa.
* Have a confirmed genetic diagnosis of Retinitis Pigmentosa secondary to mutation in the PRPF31 gene.
* For participants not previously enrolled in VP001-CL101 or VP001-CL102 studies: Meet all of the following for visual function in the study eye at the Screening Visit:

  1. Mean microperimetry threshold: >5 decibel (dB) to <15 dB
  2. Ellipsoid zone (EZ) length >1000 microns of which 500 microns is contiguous, by SD-OCT
  3. In the opinion of the Investigator, rod function is observed in any direction >10 degrees per static perimetry at Screening Visit (Visit 1)

Key Exclusion Criteria:

* Have any uncontrolled systemic disease that, in the opinion of the Investigator, would preclude participation in the study that include but are not limited to infection, uncontrolled elevated blood pressure, cardiovascular disease, or glycemic control issues, or any other medical condition that may put the participant at risk due to study procedures.
* Known mutations in genes that cause autosomal dominant RP, X-linked RP, or presence of biallelic mutations in autosomal recessive RP/retinal dystrophy genes other than PRPF31 mutations.
* Have used anti-VEGF agents within 2 months or corticosteroid injections within the last 3 months.
* Have had Ozurdex® implants placed within 3 months or Retisert® or Iluvien® implants placed within 3 years prior to Baseline (Visit 2).
* Within 3 months prior to Baseline (Visit 2), have undergone any vitreoretinal surgery or any other ocular surgery
* Have ocular media opacity or poor pupillary dilation prohibiting quality ophthalmic evaluation or photography, as assessed by the investigator.
* Have used any investigational drug or device within 90 days or 5 estimated half-lives (or within 60 days from last administration of VP-001 in the VP001-CL101 Part B or VP001-CL102 studies) of Baseline (Visit 2), whichever is longer,
* Have a recent history (<6 months) or current excessive recreational drug or alcohol use, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-03-03 (Estimated)

PRIMARY OUTCOMES:
To determine the safety of two doses of repeatedly administered intravitreally VP-001 in participants with confirmed PRPF31 mutation-associated retinal dystrophy. | 26 months
  The incidence, severity, and relatedness of ocular TEAEs and TE-SAEs in the study eye over a 26-month time period for each of the repeat doses

SECONDARY OUTCOMES:
To determine the change from Baseline (Visit 2) through End of Study/Early Termination in BCVA letter score using ETDRS charts | 24 months
  To determine the efficacy of two doses of repeatedly administered intravitreally VP-001 in participants with confirmed PRPF31 mutation-associated retinal dystrophy, RP11.
  A gain of Early Treatment Diabetic Retinopathy Study (ETDRS) letters in Best-Corrected Visual Acuity (BCVA) from Baseline through EOS/ET would indicate vision improvement.
To determine the change from baseline (Visit 2) through End of Study/Early Termination in Low Luminance Visual Acuity (LLVA) letter score | 24 months
  To determine the efficacy of two doses of repeatedly administered intravitreally VP-001 in participants with confirmed PRPF31 mutation-associated retinal dystrophy, RP11.
Change from Baseline (Visit 2) through End of Study/Early Termination in visual field sensitivity, Mean deviation (Mean Defect) as measured by standard static perimetry (Humphries) | 24 months
  To determine the efficacy of two doses of repeatedly administered intravitreally VP-001 in participants with confirmed PRPF31 mutation-associated retinal dystrophy, RP11.
Change from Baseline (Visit 2) through End of Study/Early Termination in mean retinal sensitivity | 24 months
  To determine the efficacy of two doses of repeatedly administered intravitreally VP-001 in participants with confirmed PRPF31 mutation-associated retinal dystrophy, RP11.
  > mean retinal sensitivity will be measured by fundus-guided microperimetry, measured in dB (Decibels).
Change from Baseline (Visit 2) through End of Study/Early Termination in preserved EZ area on SD-OCT | 24 months
  SD-OCT refers to Spectral Domain Optical Coherence Tomography. A preserved EZ area refers to the region of the retina where the Ellipsoid Zone (EZ), a distinct hyperreflective band representing the inner segments of photoreceptor cells, remains intact and visible, indicating relatively healthy photoreceptor function, often measured in a specific area on the scan to monitor disease progression in conditions like retinitis pigmentosa.
  To determine the efficacy of two doses of repeatedly administered intravitreally VP-001 in participants with confirmed PRPF31 mutation-associated retinal dystrophy, RP11.
Change from Baseline (Visit 2) through End of Study/Early Termination in participant reported outcome measures utilizing the Michigan Retinal Degeneration Questionnaire (MRDQ) | 24 months
  The Michigan Retinal Degeneration Questionnaire (MRDQ) is a psychometrically validated patient reported outcomes (PRO) measure for patients with inherited retinal degenerations.
  This is to determine the efficacy of two doses of repeatedly administered intravitreally VP-001 in participants with confirmed PRPF31 mutation-associated retinal dystrophy, RP11.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Florida College of Medicine, Jacksonville, Florida
  - Bascom Palmer Eye Institute - University of Miami, Miami, Florida
  - Kellogg Eye Center - University of Michigan, Ann Arbor, Michigan
  - Casey Eye Institute - OHSU, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No